CLINICAL TRIAL: NCT06589037
Title: "Comparison of Shockwave Application on the Sole of the Foot Vs. the Back of the Leg in the Treatment of Plantar Fasciitis: a Clinical Trial."
Acronym: SW-PF-BL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Paula Fernández Martín, graduate university degree, University of Alcala
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shockwave Application in PF
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis, shockwaves, sciatic nerve.
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Forty-eight subjects who meet the inclusion criteria will be recruited and randomly assigned to each intervention group. The control group will receive local shock wave therapy, while the experimental group will receive shock wave therapy along the course of the sciatic nerve.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): A group of 24 people receive shock waves along the leg to treat their plantar fasciitis.
  Interventions: Other: shock wave treatment experimental group
- Control group (Active Comparator): A group of 24 people receive shock waves on the sole of the foot to treat their plantar fasciitis
  Interventions: Other: shock wave treatment control group

INTERVENTIONS:
Other: shock wave treatment control group — The control group, consisting of 24 people, will receive shock wave treatment on the sole of the foot to treat plantar fasciitis. There will be 4 sessions and 4 data collections.
  Arms: Control group
Other: shock wave treatment experimental group — The experimental group, consisting of 24 people, will receive shockwave treatment on the back of the leg to treat plantar fasciitis. There will be 4 sessions and 4 data collections.
  Arms: experimental group

SUMMARY:
The study focuses on plantar fasciitis, one of the most common causes of non-traumatic foot and ankle pain, with an estimated prevalence of 10%. Its objective is to evaluate the effectiveness of shock wave therapy applied along the course of the sciatic nerve in treating plantar fasciitis, comparing its effects on pain, foot-ankle functionality, and quality of life.

Forty-eight subjects will be recruited and randomly assigned to two groups: one will receive local shock wave therapy, while the other will receive therapy along the sciatic nerve. Data will be collected at four points in time: before the intervention, one week after, one month after, and three months after, with blinded data collection.

Pain, foot-ankle functionality, and quality of life will be measured. Data analysis will be performed using SPSS 29.0, applying ANOVA and other tests depending on the normality of the data. Differences will be estimated with a 95% confidence interval and a p-value < 0.05.

DETAILED DESCRIPTION:
Introduction: Plantar fasciitis is one of the most common causes of non-traumatic ankle-foot pain. The exact prevalence is unknown, but it is estimated to be around 10%.

Objective: To evaluate the efficacy of applying shock waves along the course of the sciatic nerve in the treatment of plantar fasciitis and its effect on pain, as well as to assess changes in ankle-foot functionality and quality of life.

Material and Methods: Forty-eight subjects who meet the inclusion criteria will be recruited and randomly assigned to each intervention group. The control group will receive local shock wave therapy, while the experimental group will receive shock wave therapy along the course of the sciatic nerve.

Data Collection: Data will be collected at four different times: before the intervention, one week after, one month after, and three months after. The data collection will be carried out by a team member who will be blinded to the group to which the subject belongs. The dependent variables to be measured are pain (VAS scale), ankle-foot functionality (FFI), and quality of life (SF12).

Data Analysis: The data analysis will use SPSS 29.0. Normality of variables will be assessed, and descriptive analyses will be conducted. Initial homogeneity between groups will be compared, and ANOVA and other tests will be applied according to normality and homoscedasticity. Differences and percentage changes will be calculated, estimating effect size, with a 95% CI and p < .05.

ELIGIBILITY:
Inclusion criteria: having been diagnosed with plantar fasciitis, experiencing pain related to the condition for at least 1 month, and being between 18 and 65 years of age.

Exclusion criteria: being pregnant, having a pacemaker, presenting with rheumatoid arthritis, or having coagulation disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
pain (EVA scale) | 3 months
  Assess changes in pain in plantar fasciitis after treatments
ankle-foot functionality (FFI) | 3 months
  assess the improvement in ankle-foot functionality after treatment.
quality of life (SF12) | 3 months
  assess the improvement in the patient's quality of life after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernandez-Martin, Principal Investigator — University of Alcala
Locations (1):
- Campus Cientifico -Tecnológico UAH. Av. de León, 3A., Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bicer M, Hocaoglu E, Aksoy S, Inci E, Aktas I. Assessment of the Efficacy of Extracorporeal Shockwave Therapy for Plantar Fasciitis with Magnetic Resonance Imaging Findings. J Am Podiatr Med Assoc. 2018 Mar;108(2):100-105. doi: 10.7547/15-106. PMID 29634309